CLINICAL TRIAL: NCT06181825
Title: Investigating the Efficacy of a Behavioral Activation Low Intensity Intervention in Online Research Participants
Brief Title: Behavioral Activation in Depressed Online Workers
Acronym: BA-Prol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Lorenzo Lorenzo-Luaces, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19958
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Depression; Anxiety
Keywords: emotion regulation
MeSH Terms: conditions — Depression; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMET-BA (Experimental): COMET-BA (Common Elements Toolbox- Behavioral Activation) includes 4 online weekly modules which focus on elements of behavioral activation, including positive activity scheduling, avoidance reduction, values, and change plans.
  Interventions: Behavioral: COMET-BA (Common Elements Toolbox- Behavioral Activation)
- Waitlist Control (No Intervention): Thoss assigned to the waitlist control condition will complete weekly surveys but will not have access to the COMET-BA materials until the data collection period is over.

INTERVENTIONS:
Behavioral: COMET-BA (Common Elements Toolbox- Behavioral Activation) — COMET-BA includes 4 online weekly modules which focus on elements of behavioral activation, including positive activity scheduling, avoidance reduction, values, and change plans.
  Arms: COMET-BA

SUMMARY:
In this study, the investigators will test the effectiveness of a digital, low intensity mental health intervention in depressed individuals. There will be two conditions: the Common Elements Toolbox- Behavioral Activation (COMET-BA) intervention and a waiting list control group. COMET-BA will include 4 weekly modules which will focus on elements of behavioral activation, including positive activity scheduling, avoidance, values, and change plans. A similar intervention, was previously tested in an online worker sample and participant feedback was integrated into the current version of the intervention.

DETAILED DESCRIPTION:
Participants who follow the study link in Prolific will immediately be taken to the Informed Consent Statement (ICS), which will include a description of the study, risks and benefits, payment, eligibility and confidentiality. After reading the ICS, participants will confirm their consent by clicking "I consent to participate in this study." They will then be taken to the welcome page for the study and confirm that they will provide their best answers (see Attachments, "Screener"). Once participants have confirmed their consent, they will be asked screener and demographic questions (i.e., age, sex assigned at birth, gender, race/ethnicity, sexual orientation, relationship status, education level, annual income, employment status, if they have ever taken psychiatric medication/engagement in mental health services, how many people they can rely on for social support, physical health, how often they drink alcohol, and how old they were when they first struggled with depression, anxiety, or stress). In order to participate in the study, they must indicate "yes" that they are interested in learning coping skills for their mental health at this time. This is meant to address potential bias for online workers to participate in order to receive compensation without interest in adhering to the intervention if randomized to the treatment arm. Additionally, they will be administered the Patient Health Questionnaire 9-item (PHQ-9) and must reach the threshold for elevated depression symptoms (total score > 9). Information about the screener (e.g., types of questions) is provided to participants in the Informed Consent Form. Total time to complete the screener is about 3 minutes.

Participants who are ineligible will be automatically sent to a page that notifies them they do not qualify for the study. At this point their participation will be terminated.

Participants who are eligible for the study will then be prompted to complete the Week 1 Questionnaire (see Attachments, "Week 1") via the Prolific platform. Study team will send out a Bulk Message to eligible participants to complete the weekly modules on a week-by-week basis. The message to participants can be found in the Attachments, "Message". In this questionnaire they will fill out a series of measures including: the Generalized Anxiety Disorder 7-item (GAD-7), WHO-5 Well-being Index (WHO-5), 3 questions from the Insomnia Severity Index (ISI), Emotion Regulation Questionnaire (ERQ), Ten-Item Personality Inventory (TIPI), Adverse Childhood Experiences Scale (ACES), Work and Social Adjustment Scale (WSAS), and the Behavioral Activation for Depression Scale Activation Subscale (BADS-AC). After completing these questionnaires participants will be randomized to either the COMET-BA intervention condition or the control condition (which will receive access to the intervention after 8 weeks ). This randomization will be completed via the Qualtrics randomizer function - which randomly and evenly assigns participants to the two conditions.

Participants who are assigned to the COMET-BA condition will then be taken to the first intervention module (see Attachments, "Week 1"). They will then receive the first module, Positive Activity Scheduling, where participants will learn about the theory underlying behavioral activation and impact of scheduling positive activities. They will be asked to brainstorm and plan a positive activity they can do in the next week. In total, the time estimate for week 1 is about 10 minutes. Participants in the control condition will be notified of the condition assignment and reminded about upcoming weekly questionnaires but will not receive the module for week 1 until the study is over. The time to complete Week 1 for the control condition is about 5 minutes.

In the next week, participants will have access to the Week 2 modules through the Prolific platform and sent a message through the Prolific platform (see attachments "Message"). All participants will complete the weekly outcome measures, including the GAD-7, PHQ-9, WHO-5, ERQ, WSAS, and BADS-AC. For those in the COMET-BA condition, they will receive the Avoidance module (see Attachments, "Week 2"). First, participants will complete the weekly outcome measures, including the GAD-7, PHQ-9, WHO-5, ERQ, WSAS, and BADS-AC. Participants in the COMET-BA condition will then be asked about their adherence to last week's plan, receive psychoeducation around the nature of avoidance in depression, and complete an exercise to practice identifying avoidance strategies before they complete the another positive activity scheduling exercise for the upcoming week. In total, the time estimate for week 2 is about 10 minutes. Participants in the control condition will be administered the questionnaires alone and not the COMET-BA module. The time to complete the questionnaires for Week 2 is about 5 minutes.

In the third week, participants will have access to the Week 3 modules through the Prolific platform and sent a message through the Prolific platform (see attachments "Message"). Participants will complete the weekly outcome measures, including the GAD-7, PHQ-9, WHO-5, ERQ, WSAS, and BADS-AC, and then have access to the Week 3 modules through the Prolific platform. For those in the COMET-BA condition, they will receive the Values module (see Attachments, "Week 3"). First, participants will complete the weekly outcome measures, including the GAD-7, PHQ-9, WHO-5, ERQ, WSAS, and BADS-AC. Participants in this module will again be asked about their adherence to last week's plan, receive psychoeducation around the nature of and benefit to acting on one's values, and complete an exercise to practice identifying their values and a plan to act on them in the upcoming week. In total, the time estimate for Week 3 is about 10 minutes. Participants in the control condition will be administered the questionnaires alone and not the COMET-BA module. The time to complete the questionnaires for Week 3 is about 5 minutes.

In the fourth week, participants will have access to the Week 4 modules through the Prolific platform and sent a message through the Prolific platform (see attachments "Message"). Participants will complete the weekly outcome measures, including the GAD-7, PHQ-9, WHO-5, ERQ, WSAS, and BADS-AC, and then have access to have access to the Week 4 modules through the Prolific platform. For those in the COMET-BA condition, they will receive the Change Plan module (see Attachments, "Week 4"). First, participants will complete the weekly outcome measures, including the GAD-7, PHQ-9, WHO-5, ERQ, WSAS, and BADS-AC. Participants in this module will again be asked about their adherence to last week's plan, then receive psychoeducation around the nature of change plans and complete a change plan exercise for the future. In total, the time estimate for Week 4 is about 10 minutes. Participants in the control condition will be administered the questionnaires alone and not the COMET-BA module. The time to complete the questionnaires for Week 4 is about 5 minutes.

Participants who are assigned to the control condition will receive weekly links through Prolific similar to the COMET-BA condition, but rather than receiving a module they will be directed to a series of questionnaires identical to the weekly questionnaires outlined in the COMET-BA condition (GAD-7, PHQ-9, WHO-5, ERQ, WSAS, and BADS-AC). This is all the control condition will be completing. Provided the intervention condition will entail completing an online, survey-style intervention, the control condition will similarly be completing weekly surveys as a "waitlist" condition until the end of the study, when the intervention materials will be made available freely for all participants. All surveys and intervention materials will end with a mental wellbeing resource list (see Attachments, "Resource List") for both the Control and COMET-BA groups.

After completing the COMET-BA intervention, all participants from both conditions will receive a 1-week follow-up after the completion of the Week 4 module (see Attachments, "Follow-Up 1"). This will include the PHQ-9, GAD-7, WHO-5, ERQ, ISI, WSAS, and the BADS-AC. The same questionnaire will be sent out 3 weeks later to establish a 4-week follow-up (see Attachments, "Follow-Up 2"). Thus, the total time for the study from start to end is about 8 weeks. In the informed consent statement, participants will be informed that there are follow-up assessments that they can receive additional compensation for. The study team will also put a message at the end of each module reminding them to watch for the follow ups. They will not be notified of these follow-up assessments, but will be able to see the follow-up assessments posted on Prolific. Participants who do not complete the follow up assessments within 1 day will be sent a reminder within Prolific's system (see Attachments, "COMET-BA Prolific Follow Up Reminder"). During these follow-ups all participants (e.g., those in both the intervention and control conditions) will complete the following questionnaires: GAD-7, PHQ-9, WHO-5, ISI, ERQ, WSAS, and BADS-AC.

After completing the follow-up measure at 8 weeks, enrollment in the study will end. At this point, participants in the control condition will receive the intervention modules via a link through the Prolific platform (see "Final Message Prolific"). Whether they complete the intervention or not is entirely up to them and it will not be tracked by the research team. Their use of the COMET intervention is entirely optional and will not be recorded by the research team. They will not fill out any follow up measures after completing or not completing the COMET intervention. The materials are made available so they may also access the materials available to those in the intervention condition as they may desire.

ELIGIBILITY:
Inclusion Criteria:

* PHQ9 > 9 at baseline, indicate "yes" that they are interested in learning coping skills for their mental health

Exclusion Criteria:

* PHQ9 < or = 9 at baseline, indicate they are not interested in learning coping skills for mental health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | 8 weeks
  Depression symptoms will be assessed with the PHQ-9. The PHQ-9 is a 9-item self-report measure that assesses the frequency of symptoms of major depressive disorder as outlined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Response options range from 0 ("not at all") to 3 (nearly every day). Total scores on the PHQ-9 range from 0-27 with greater scores indicating greater frequency of depressive symptoms. A score greater than or equal to 10 on the PHQ-9 has been identified as a positive screen for major depression (Kroenke & Spitzer, 2002). PHQ-9 will be assessed at baseline, each week of the intervention, and 1-week and 4-weeks post-intervention follow-up.
Generalized Anxiety Disorder Scale-7 (GAD-7) | 8 weeks
  Anxiety symptoms will be assessed with the GAD-7, a 7-item self-report measure that assesses the frequency of anxiety symptoms. Responses range from 0 ("not at all") to 3 ("nearly every day"), yielding total scores that range from 0-21 with greater scores indicating greater frequency of anxiety symptoms. A score greater than or equal to 10 on the GAD-7 has been identified as a positive screen for anxiety in primary care settings (Spitzer et al., 2006). GAD-7 will be assessed at baseline, each week of the intervention, and 1-week and 4-weeks post-intervention follow-up.
World Health Organization Well-Being Index-5 (WHO-5) | 8 weeks
  Well-being will be assessed with the WHO-5, a 5-item self-report measure of subjective well-being. Items are rated on a 6-point Likert scale ranging from 0 ("at no time") to 5 ("all of the time"), yielding total raw scores that range from 0-25. Raw scores are multiplied by four to generate a score from 0-100 with greater scores indicating higher levels of subjective well-being. A score of 50 is considered the cutoff to screen for major depression (Topp et al., 2015). WHO-5 will be assessed at baseline, each week of the intervention, and 1-week and 4-weeks post-intervention follow-up.

SECONDARY OUTCOMES:
Emotion Regulation Scale (ERQ) | 8 weeks
  The ERQ (Gross & John, 2003) is a ten-item self-report measure of individual differences in the use of two emotion regulation strategies: cognitive reappraisal (ERQ-reappraisal; items 1, 3, 5, 6, 8, and 10) and expressive suppression (ERQ-suppression; items 2, 4, 6, and 9). The ERQ items are rated on a seven-point Likert scale with responses ranging from 1 ("strongly disagree") to 7 ("strongly agree"). The research team will average item scores to produce final scores on the same metric of the original items (i.e., 1 to 7) in order to make the ERQ-reappraisal and ERQ-suppression subscales (with differing numbers of items) comparable. The ERQ will be assessed at baseline, each week of the intervention, and 1-week and 4-weeks post-intervention follow-up.
Behavioral Activation for Depression Scale Activation Subscale (BADS-AC) | 8 weeks
  The BADS is a self-report questionaire of behavioral activation that consists of 25 questions, each rated on a seven-point scale ranging from 0 ("not at all") to 6 ("completely"). The Activation subscale consists of 10 of the questions in the BADS. Items from the Activation subscale are summed to yield a total score of 0-60, with greater scores indicating greater activation. The BADS-AC will be assessed at baseline, each week of the intervention, and 1-week and 4-weeks post-intervention follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peipert A, Lorenzo-Luaces L. Is there a treatment for the Turker blues? A fully remote nationwide randomized controlled trial of a digital intervention for depression in adult online workers. J Consult Clin Psychol. 2025 Nov;93(11):719-734. doi: 10.1037/ccp0000982. PMID 41182705